CLINICAL TRIAL: NCT06799260
Title: Priming Effects of Ketone Monoester Supplementation on Theta-Burst Stimulation-Induced Plasticity in the Primary Motor Cortex
Brief Title: Motor Cortex Plasticity Response to Theta-Burst Stimulation After Ketone Monoester Supplementation
Acronym: KME-TBS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, Wan Aliaa Wan Sulaiman, Associate Professor, Universiti Putra Malaysia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: JKEUPM-2021-485; FRGS/1/2022/SKK01/UPM/02/4 (Other Grant/Funding Number: Ministry of Higher Education, Malaysia)
Record Dates: First submitted 2025-01-02; First posted 2025-01-29 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-12

CONDITIONS: Healthy Young Adult; Neurophysiology
Keywords: Transcranial magnetic stimulation; Intermittent theta-burst stimulation; Continuous theta-burst stimulation; Primary motor cortex; Neuroplasticity; ketone monoester; Beta-hydroxybutyrate; Brain-derived neurotrophic factor; Blood pressure; Heart rate

STUDY DESIGN:
Intervention Model Description: This is a partial crossover study.
  The study protocol involves two interventions administered sequentially during each visit:
  Supplement intervention (KME/placebo) followed after one hour by a stimulation intervention (iTBS/cTBS).
  There will be two separate groups of subjects undergoing different TBS protocols (iTBS vs cTBS).
  The subjects of each group will crossover the supplement intervention (KME and placebo) in two visits separated by one week.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- KME then placebo supplement with iTBS stimulation (Experimental): KME drink with iTBS stimulation over the left M1 hand region, followed after a 1-week washout period by a placebo drink with iTBS stimulation over the left M1 hand region
  Interventions: Dietary Supplement: Ketone Monoester (KME); Dietary Supplement: Placebo; Device: iTBS
- Placebo then KME supplement with iTBS stimulation (Experimental): Placebo drink with iTBS stimulation over the left M1 hand region, followed after a 1-week washout period by a KME drink with iTBS stimulation over the left M1 hand region
  Interventions: Dietary Supplement: Ketone Monoester (KME); Dietary Supplement: Placebo; Device: iTBS
- KME then placebo supplement with cTBS stimulation (Experimental): KME drink with cTBS stimulation over the left M1 hand region, followed after a 1-week washout period by a placebo drink with cTBS stimulation over the left M1 hand region
  Interventions: Dietary Supplement: Ketone Monoester (KME); Dietary Supplement: Placebo; Device: cTBS
- Placebo then KME supplement with cTBS stimulation (Experimental): Placebo drink with cTBS stimulation over the left M1 hand region, followed after a 1-week washout period by a KME drink with cTBS stimulation over the left M1 hand region
  Interventions: Dietary Supplement: Ketone Monoester (KME); Dietary Supplement: Placebo; Device: cTBS

INTERVENTIONS:
Dietary Supplement: Ketone Monoester (KME) — 500 mg/kg body weight of the KME supplement
Dietary Supplement: Placebo — Taste-matched placebo drink
Device: iTBS — iTBS stimulation will be applied using a butterfly figure-of-eight Cool-B70 coil connected to a MagPro R30 stimulator with add-on Theta Burst option (MagVenture A/S, Farum, Denmark).
  Arms: KME then placebo supplement with iTBS stimulation; Placebo then KME supplement with iTBS stimulation
Device: cTBS — cTBS stimulation will be applied using a butterfly figure-of-eight Cool-B70 coil connected to a MagPro R30 stimulator with add-on Theta Burst option (MagVenture A/S, Farum, Denmark).
  Arms: KME then placebo supplement with cTBS stimulation; Placebo then KME supplement with cTBS stimulation

SUMMARY:
Transcranial magnetic stimulation is a medical device that can alter motor cortical (M1) excitability through the scalp via various protocols. Among these, intermittent- and continuous-theta burst stimulation (iTBS/cTBS) are increasingly used protocols to enhance or suppress M1 excitability, respectively, beyond stimulation. However, the poor reproducibility and high inter-individual variability in responses to TBS protocols are matters of concern. This study will explore whether ketone monoester supplementation can boost TBS efficacy via their mechanistic convergence on Brain-Derived Neurotrophic Factor (BDNF).

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adults (18-35 years old)
* Right-handed
* Fully vaccinated against COVID-19

Exclusion Criteria:

* Subjects with contraindications to TMS based on the screening 13-item questionnaire for TMS safety
* Highly active subjects (athletes)
* Obese (BMI ≥ 30 kg/m2)
* Smokers
* Following intermittent fasting or ketogenic diet
* Long COVID-19

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Motor evoked potential (MEP) | Pre-TBS (baseline) and post-TBS at 0, 5, 10, 20, and 30 minutes.
  Peak-to-peak MEP amplitude elicited by single-pulse TMS over the left M1 representation of the first dorsal interosseous (FDI) muscle.
  In each MEP measurement, 12 MEP readings will be collected, elicited by single-pulse TMS at an intensity of 120% resting motor threshold and separated by 15 seconds.
  In each timepoint post-TBS, the mean value of MEPs (aka, conditioned MEPs) will be averaged and compared to pre-TBS (aka, baseline MEPs) using the following equation: (conditioned MEP amplitude/baseline MEP amplitude) × 100. A value of 90-110 represents no change, while values < 90% represent suppression and > 110% facilitation of the M1 plasticity following TBS.

SECONDARY OUTCOMES:
TMSens_Q questionnaire | At 30 minutes post-TBS stimulation
  Self-reported side effects using the TMSens_Q questionnaire to evaluate the tolerability of the KME-TBS combination.
Corticospinal excitability indices | Pre-KME supplementation and at 1 hour post-KME supplementation
  Resting motor threshold (RMT) followed by motor-evoked potential at 120% RMT intensity
Blood pressure | Pre-supplementation, at 1 hour post-supplementation/pre-TBS stimulation, and serially thereafter every 3-5 minutes until 30 minutes post-TBS
  Systolic blood pressure (SBP), Diastolic Blood Pressure (DBP), and Mean Arterial Pressure (MAP) using fully automated oscillometric sphygmomanometer
Heart rate | Pre-supplementation, at 1 hour post-supplementation/pre-TBS stimulation, and continuously thereafter for 30 minutes post-TBS
  Heart rate (bpm) using pulse oximeter
Blood glucose | Pre-KME supplementation and at 30 minutes post-TBS stimulation
  On-site using a portable glucometer
Blood beta-hydroxybutyrate | Pre-KME supplementation and at 30 minutes post-TBS stimulation
  On-site using a portable glucometer
Serum brain-derived neurotrophic factor | Pre-KME supplementation and at 30 minutes post-TBS stimulation
  Serum levels of mature brain-derived neurotrophic factor (mBDNF) and pro-BDNF isoforms
BDNF genetic polymorphism | At the baseline (pre-KME supplementation)
  BDNF rs6265 single nucleotide polymorphism

CONTACTS AND LOCATIONS:
Overall Officials: Wan Aliaa Wan Sulaiman, FRCP, Study Chair — Universiti Putra Malaysia
Locations (1):
- Hospital Sultan Abdul Aziz Shah, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified raw datasets collected during the trial will be freely available upon completion on the Open Science Framework repository at https://osf.io/
URL: https://osf.io/